CLINICAL TRIAL: NCT03398226
Title: Chronological Change of Bone Microstructure After Gastrectomy
Brief Title: Bone Microstructure After Gastrectomy Evaluating by Using HR-pQCT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nagasaki University (Other)
Responsible Party: Principal Investigator, Kobayashi Shinichiro, Principal Investigator in department of Surgery, Nagasaki University
Other Study IDs: 17082126
Record Dates: First submitted 2017-09-17; First posted 2018-01-12 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Osteoporosis; Sarcopenia; Gastric Cancer
MeSH Terms: conditions — Osteoporosis; Sarcopenia; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group
- Distal Gastrectomy (DG) group: 38 patients planing distal gastrectomy due to gastric cancer
- Total Gastrectomy (TG) group: 38 patients planing total gastrectomy due to gastric cancer

SUMMARY:
Osteoporosis after gastrectomy, which is characterized by both the loss of bone mass and the deterioration of bone architecture, is a serious complication in the long course after gastrectomy. The aim of the present study was to evaluate osteoporosis by using high-resolution peripheral quantitative computed tomography (HR-pQCT) in the long course after gastrectomy. In total gastrectomy and distal gastrectomy groups, at least 5 years should have elapsed since gastrectomy.

DETAILED DESCRIPTION:
The patients after gastrectomy loss appetite and decrease the weight. Total gastrectomy especially cause severe sarcopenia and metabolic change. Osteoporosis after gastrectomy, which is characterized by both the loss of bone mass and the deterioration of bone architecture, is a serious complication in the long course after gastrectomy. The primary tools for assessing volumetric density and bone structure are quantitative computed tomography (QCT) and more recently, high-resolution peripheral quantitative computed tomography (HR-pQCT). However the validation of osteoporosis with HR-pQCT before and after gastrectomy remain elusive. The aim of the present study was to evaluate osteoporosis by using HR-pQCT before and after after endoscopic resection, distal gastrectomy, and total gastrectomy in the patients with gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Planning ESD, DG, or TG due to gastric cancer
* Provide signed informed consent

Exclusion Criteria:

* pregnancy
* Current use of the following osteoporosis agents; Teriparatide, Denosumab, and bisphosphonate
* Hyperthyroidism
* Hyperparathyroidism
* Present malignancy (except in situ carcinoma)
* Any condition that required chronic (greater than three months cumulative and greater than 5 mg/day) glucocorticoid therapy
* Other diseases which affect bone metabolism
* Any disorder that, in the opinion of the investigator, may compromise the ability of the subject to give written informed consent and/or comply with study procedures
* Received > 3 months (or equivalent) of osteoporosis treatment
* Currently enrolled in or has not yet completed at least 1 month since ending other investigational device or drug trial(s), or subject is receiving other investigational agent(s).

Ages: 60 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Japanese
Sampling Method: Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2017-09-18 (Actual); Primary Completion 2020-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Comparing bone microstructure in control, DG, and TG groups | 2 years after the treatments
  volumetric bone mineral density loss comparing with before the treatments

SECONDARY OUTCOMES:
Comparing bone microstructure with sarcopenia | Before the treatments and 1 and 2 years after the treatments
  Correlation between bone mineral density in HR-pQCT and cross-sectional area of the abdominal psoas major muscle
Comparing bone microstructure with serum biomarkers of osteoporosis | Before the treatments and 1 and 2 years after the treatments
  Correlation between bone mineral density in HR-pQCT and biomarkers (25-hydroxyvitaminD, calcium, iPTH, P1NP, ICTP, TRACP5b)
Comparing bone microstructure with dual-energy X-ray absorptiometry | Before the treatments and 1 and 2 years after the treatments
  Correlation of bone mineral density between HR-pQCT and DXA
Comparing bone microstructure with quality of life (QOL-C30) | Before the treatments and 1 and 2 years after the treatments
  Patients will be asked to complete a short debriefing questionnaire covering questions.(QOL-C30). We compared the average sore about Valid and reliable 30-item questionnaire assessing health related quality of life (6 functional, 9 symptom) before and after treatments. The score about QOL-C30 is evaluated on a four level scale without Global quality of life. Global quality of life is evaluated on a seven level scale.
Comparing bone microstructure with quality of life (BDHQ) | Before the treatments and 1 and 2 years after the treatments
  Patients will be asked to complete a short debriefing questionnaire covering questions (BDHQ) B-DHQ is 58-item fixed-portion-type questionnaire The score about BDHQ is evaluated on a seven level scale.
Comparing bone microstructure with quality of life (FRAX) | Before the treatments and 1 and 2 years after the treatments
  Patients will be asked to complete a short debriefing questionnaire covering questions (FRAX). FRAX score is 12. FRAX is 12-item fixed-portion-type questionnaire. The score about FRAX is evaluated on a two level scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Nagasaki University Hospital, Nagasaki, Japan

IPD SHARING:
Plan to Share IPD: No